CLINICAL TRIAL: NCT06523179
Title: Study for the Evaluation of Risk of hEpatocellular Carcinoma in NonAlcoholic Fatty Liver
Brief Title: Evaluation of Risk of hEpatocellular Carcinoma
Acronym: PERSPECTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Valenti:, Clinical Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PERSPECTIVE
Record Dates: First submitted 2024-03-07; First posted 2024-07-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: NASH; HCC; Genetic Predisposition
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk factors for NAFLD-HCC (Experimental): The study will be divided into:
  * In the first phase, the impact of a score based on the evaluation of common genetic variants in genes predisposing to the development of NAFLD-HCC (PNPLA3, TM6SF2, and MBOAT7), and rare mutations determining high risk of NAFLD-HCC, e.g. . in genes involved in telomere shortening (TERT) and lipid metabolism (APOB) on the risk of developing HCC and on survival, in the entire cohort of patients and in the individual groups listed above.
  * In the second phase we will use next generation sequencing techniques (whole exome / genome sequencing) to identify new genetic risk variants for the development of HCC.
  Interventions: Other: quantify the impact of genetic risk factors

INTERVENTIONS:
Other: quantify the impact of genetic risk factors — the impact of genetic risk factors for the development of NAFLD-HCC and their interaction with acquired risk factors, on the incidence of the disease in a prospective cohort of patients at risk, through a score capable of predicting NAFLD-HCC and selecting patients for whom screening is cost-effective.

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common solid cancer and the second cause of cancer-related mortality worldwide. Nonalcoholic fatty liver disease (NAFLD), that is hepatic accumulation of fat in excess of 5% not explained by at risk alcohol intake, is projected to become the leading cause of HCC in Western countries within 2025.NAFLD is most frequently caused by insulin resistance due to unhealthy lifestyle. Due to the epidemics of obesity and type 2 diabetes, NAFLD now affects one in three individuals worldwide.

NAFLD-HCC frequently develops without overt cirrhosis suggesting that steatosis directly promotes hepatic carcinogenesis.

DETAILED DESCRIPTION:
The mechanisms linking NAFLD to liver disease progression towards HCC have not yet been identified. Anyhow several pathways may be activated in obesity and diabetes favoring a tumor-promoting environment distinguishing the pathogenesis of NAFLD-HCC from that of other etiologies. First of all, increased cancer risk is associated with a low-grade of chronic inflammation, a manifestation typical of obesity and metabolic syndrome. Indeed, adipose tissue expansion promotes the release of pro-inflammatory cytokines, namely tumor necrosis factor alpha (TNFα) and interleukin 6 (IL6) both potent activators of key oncogenic signaling pathways. Furthermore, obesity alters the release of adipokines reducing the level of those with anti-inflammatory effects such as adiponectin and arising the level of those with pro-inflammatory and fibrogenic effects, such as leptin. Overall the factors listed above collectively induce hyperinsulinemia, resulting in increased bioavailability of insulin-like growth factor-1 (IGF1) which in turn promotes cellular proliferation and inhibits apoptosis. The activation of hepatic stellate cells (HSCs) is also a major step in the development of cirrhotic HCC, however these cells not only secrete collagen that results in liver fibrosis, but may even produce several growth factors which stimulate oncogenic pathways contributing to the expansion of neoplastic clones.

Genetic factors have been shown to influence disease progression in NAFLD, and family history remains the main risk factor for HCC development. The common genetic polymorphism rs738409 C>G encoding for the I148M variant in Patatin-like phospholipase domain-containing protein 3 (PNPLA3 or adiponutrin) has been established as the main common genetic determinant of hepatic fat content and of progressive NAFLD. The mechanism is related to accumulation of the mutated protein, which interferes with lipid droplets remodeling in hepatocytes, and with retinol release by hepatic stellate cells. The PNPLA3 variant predicts HCC development in European patients with NAFLD. This evidence suggests that this genetic risk factors may be helpful to select high-risk individuals for screening, but it has a low sensitivity to be used as single prognostic biomarker. The rs58542926 E167K variant in Transmembrane 6 superfamily member 2 (TM6SF2) also predisposes to progressive NAFLD by altering the secretion of very low-density lipoproteins, but its direct role in HCC predisposition is disputed. More recently, it has been found that the rs641738 C>T sequence variant in the Membrane bound O-acyltranferase domain containing 7/ Transmembrane channel like 4 (MBOAT7/TMC4) locus, involved in phospholipids remodeling, predisposes to cirrhosis development in individuals with excessive alcohol intake, and to the development and the progression of NAFLD in individuals of European descent. We recently reported in a cross sectional cohort that the rs641738 variant is also associated with HCC risk is patients with NAFLD .

Moreover, loss of function germline mutations in the telomerase reverse transcriptase (hTERT) can predispose to a spectrum of familial liver diseases characterized by steatosis and possible evolution to cirrhosis and HCC. Furthermore, it has also been reported that rare mutations inducing Mendelian diseases due to severe derangements in the function of encoded proteins may predispose to NAFLD-HCC. Indeed, mutations in Apolipoprotein B (APOB) may explain some familial cases through predisposition towards development of severe steatosis caused by hepatocellular retention of lipids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD or cryptogenic liver disease, allowing a more liberal alcohol intake limit (<60/40 g/day in M/F), so as to also include subjects with a moderate alcoholic component of liver disease, an important factor given the high epidemiological burden of this group
* Age between 45 and 75 years
* Any of the following criteria:
* F3-F4 fibrosis, determined histologically, or by non-invasive techniques (stiffness > 7.9 kPa at Fibroscan and positivity at the NAFLD fibrosis score or at APRI or at FIB4), or evidence of cirrhosis deriving from biochemical tests or imaging methods;
* Family history of primary liver cancer in first degree parentage, or carrier status of rare mutations associated with the development of HCC (such as mutations in APOB and TERT)
* Male patient with type 2 diabetes or obesity carrying at least three genetic variants in PNPLA3, TM6SF2, MBOAT7.
* Willingness to sign the informed consent.

Exclusion Criteria:

* Alcohol intake >60/40 g/day in M/F
* Chronic viral or autoimmune hepatitis
* Any previously diagnosed genetic liver disease associated with increased risk of HCC (such as hereditary hemochromatosis, Wilson's disease, Alpha-1 Antitrypsin deficiency)
* Use of drugs known to induce steatosis and liver disease
* HCC diagnosed before the study start date.
* Other pathological conditions with a prognosis of less than two years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
The quantify the impact of genetic risk factors for NAFLD-HCC and their interaction | up to 84 months
  The different inclusion criteria are able to identify the number of individuals at risk for NAFLD-HCC among patients with NAFLD following up, Understand the impact of individual genetic variants on HCC risk and rates of patients hosting gene mutations in evolving fat accumulation in liver (global cohorts and according to enrolment criteria)
The quantify the impact of genetic risk factors for NAFLD-HCC and their interaction | up to 84 months
  The impact of genetic risk factors for NAFLD-HCC and their interaction will be realized by evaluating the interaction with risk factors and developing a score to predict NAFLD-HCC. These elements will enable us to select patients for whom screening can be effective.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT06523179/Prot_SAP_000.pdf